CLINICAL TRIAL: NCT01242553
Title: Clinical Validation Study for iVue
Status: Completed | Type: Observational
Sponsor: Optovue (Industry)
Responsible Party: Director of Clinical Affairs, Optovue
Other Study IDs: iVue 100-2009
Record Dates: First submitted 2010-11-15; First posted 2010-11-17 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2010-11

CONDITIONS: Normal and Ocular Pathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Normal: Normal results from clinical exam and free of ocular pathology.
- Retina: Clinical exam results consistent with retina pathology
- Glaucoma: Clinical exam results consistent with glaucoma and visual field defects consistent with glaucoma.
- Cornea: Clinical exam results consistent with cornea pathology.

SUMMARY:
To demonstrate clinical substantial equivalence of iVue as comparable to commercially available RTVue.

ELIGIBILITY:
Inclusion Criteria:

* Normal: Normal results from clinical exam and free of ocular pathology.
* Glaucoma: Clinical exam results consistent with glaucoma and visual field defects consistent with glaucoma.
* Cornea: Clinical exam results consistent with cornea pathology.
* Retina: Clinical exam results consistent with retina pathology

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers with various ocular pathology or no ocular pathology.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
thickness of ocular structures

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hee, MD, Principal Investigator — Pacific Eye Specialists; Nalin Mehta, MD, Principal Investigator — Colorado Retina Center; Michael Sinai, PhD, Study Director — Optovue
Locations (2):
- United States (2):
  - Pacific Eye Specialists, Daly City, California
  - Colorado Retina Center, Denver, Colorado